CLINICAL TRIAL: NCT02897531
Title: A Comparison of Surgical Outcomes Between End-to-side and Side-to-side Anastomosis After Laparoscopic Right Hemicolectomy: A Prospective Randomized Controlled Trial
Brief Title: Comparison Between End-to-side and Side-to-side Anastomosis After Laparoscopic Right Hemicolectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung-Bum Kang, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1607-354-004
Record Dates: First submitted 2016-09-02; First posted 2016-09-13 (Estimated); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Anastomosis
Keywords: Ileocolic, stapled, laparoscopy, right hemicolectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ES anastomosis (Active Comparator): Stapled end-to-side anastomosis
  Interventions: Procedure: ES anastomosis
- SS anastomosis (Active Comparator): Stapled side-to-side anastomosis
  Interventions: Procedure: SS anastomosis

INTERVENTIONS:
Procedure: ES anastomosis — The side wall of the transverse colon will be anastomosed to the end of the distal ileum with one circular stapler, and the blind end of the transverse colon will be closed with one linear stapler.
  Arms: ES anastomosis
Procedure: SS anastomosis — The side wall of the transverse colon will be anastomosed to the side wall of the distal ileum with two linear staplers.
  Arms: SS anastomosis

SUMMARY:
The purpose of this study is to evaluate the efficacy of end-to-side anastomosis after laparoscopic right hemicolectomy compared with that of side-to-side anastomosis. The investigators hypothesize that the end-to-side anastomosis may be associated with superior recovery compared with side-to-side anastomosis after laparoscopic right hemicolectomy under enhanced recovery program. The primary endpoint is the cumulative recovery rate, consisting of the recovery time of diet, pain, ambulation, and afebrile status.

DETAILED DESCRIPTION:
All patients will be received a laparoscopic right hemicolectomy by three experienced colorectal surgeons and randomly divided into two groups according to the method of anastomosis: - the end-to-side anastomosis group and the side-to-side anastomosis group. After the surgery, enhanced recovery program will be implemented. The primary endpoint is the cumulative recovery rate according to the method of anastomosis. The cumulative recovery rate is defined as the percentage of patients who are satisfied with all aspects of recovery time, including i) tolerance of diet for 24 hours, 2) analgesic-free (oral or intravenous (IV) analgesic drugs not necessary after cessation of patient-controlled analgesia (PCA)), 3) safe ambulation (ambulation of 600m without assistance), 4) afebrile status without major complications (fever was defined as body temperature greater than 37.2°C at axilla). Secondary endpoints are postoperative hospital stay, complications, the failure rate of the enhanced recovery program, and the readmission rate within 1 month after surgery. The expected cumulative recovery rate in postoperative day 7 is 90% in the end-to-side anastomosis group and 70% in the side-to-side anastomosis group. The sample size of 130 patients was calculated as follow: Based on the assumption that cumulative recovery rate will increase to 20% using the end-to-side anastomosis, it was calculated that 65 patients should be in each group. The sample size was calculated by the formula for a power 80%, alpha error of 0.05 and dropout rate of 10%.

ELIGIBILITY:
Inclusion Criteria: Patients who have all of the following:

* Age: 18 - 80
* Right-sided colon cancer (adenocarcinoma, located in cecum to hepatic flexure)
* Appropriate laboratory (Bone marrow) findings (Hemoglobin ≥ 10g/dl, White blood cell count ≥ 4,000/mm3, Platelet ≥ 100,000/mm3)
* Appropriate renal function (Creatinine ≤ 1.5 mg/dl)
* Appropriate cardio-pulmonary functions
* Appropriate understanding of the study and provide the informed consent

Exclusion Criteria: Patients who have 1 or more of the following:

* Distant metastasis or locally advanced tumor which required combined resection of other organs, such as the ureter, duodenum, or small bowel.
* Not suitable for laparoscopic surgery
* Currently taking medication for dyschezia, such as constipation or diarrhea.
* Not suitable for adapting enhanced recovery program due to underlying diseases, such as cardio-pulmonary disease, mental disorder, and etc.
* Not suitable for participation in this clinical trial based on the judgment of the investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bum Kang, M.D, Ph.D., Principal Investigator — Seoul National University College of Medicine Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National Univercity Bundang Hospital, Seongnam, Gyeonggido
  - Seoul National University Bundang Hospital, Seongnam

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the study period, 201 patients met the inclusion criteria. Excluding patients who required combined operations (n = 18), and patients who could not undergo laparoscopic surgery or an ERAS protocol due to previous medical/surgical history (n = 22), 161 patients were invited to participate in the study. Of these, 130 provided informed consent and were randomized to either the ES or the SS group (n = 65 each)
Period: Overall Study
Arm/Group | ES Anastomosis | SS Anastomosis
Started | 65 | 65
Completed | 65 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ES Anastomosis | SS Anastomosis | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.6) | 59.7 (11.5) | 62.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 32 | 74
  Male | 23 | 33 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 65 | 65 | 130
American Society of Anesthesiology [Number; unit: participants] — the ASA score means ASA 1: A healthy patient with minimal risk ASA 2: A patient with mild systemic disease ASA 3: A patient with severe systemic disease ASA 4: A patient with severe systemic disease that is a constant threat to life ASA 5: A moribund patient who is not expected to live 24 hours with or without surgery ASA 6: A brain-dead patient with plans for organ donation
  participants
    ASA 1 | 18 | 22 | 40
    ASA 2 | 39 | 33 | 72
    ASA 3 | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Recovery Rate
Description: The cumulative recovery rate is defined as the percentage of patients who are satisfied with all aspects of recovery time. Recovery time includes the following:
  1. Tolerance of diet for 24hours
  2. Analgesic-free status (oral or intravenous (IV) analgesic drugs not necessary after cessation of patient-controlled analgesia (PCA)),
  3. Safe ambulation (ambulation of 600m without assistance),
  4. Afebrile status without major complications (fever was defined as body temperature greater than 37.2°C at axilla).
Time Frame: at 7 days after operation
Measure: Number; unit: percentage of participants
Arm/Group | ES Anastomosis | SS Anastomosis
Number analyzed (Participants) | 65 | 65
percentage of participants | 100 | 100

2. Secondary Outcome: Postoperative Hospital Stay
Description: Time(days) from operation to discharge
Time Frame: at discharge from hospital, an average of 1 week
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ES Anastomosis | SS Anastomosis
Number analyzed (Participants) | 65 | 65
days | 5 [5 to 7] | 6 [5 to 7]

3. Secondary Outcome: Postoperative Complications
Description: Includes any minor complication (ileus, wound infection) to major complications requiring re-intervention
Time Frame: at 30 days
Measure: Number; unit: events
Arm/Group | ES Anastomosis | SS Anastomosis
Number analyzed (Participants) | 65 | 65
events | 11 | 8

4. Secondary Outcome: Failure Rate of the Enhanced Recovery Program
Description: the number of patients who failed to adhere to the ERAS protocol
Time Frame: at discharge from hospital, an average of 1 week
Measure: Number; unit: participants
Arm/Group | ES Anastomosis | SS Anastomosis
Number analyzed (Participants) | 65 | 65
participants | 7 | 5

5. Secondary Outcome: Readmission Rate Within 1 Month After Surgery
Description: the number of patients who were re-admitted after discharge within 1 month after surgery
Time Frame: at 30 days
Measure: Number; unit: participants
Arm/Group | ES Anastomosis | SS Anastomosis
Number analyzed (Participants) | 65 | 65
participants | 3 | 2

ADVERSE EVENTS:
Time Frame: up to 3 year for each participant
Arm/Group | ES Anastomosis | SS Anastomosis
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 8/65 | 6/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ES Anastomosis (N=65) | SS Anastomosis (N=65)
ileus (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Surgical site infection (Infections and infestations) | 5 (5) | 3 (3)

LIMITATIONS AND CAVEATS:
Second, our ERAS protocol did not include recent developments such as preoperative carbohydrate loading, multimodal analgesia, and routine administration of drugs for prevention of postoperative nausea and vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT02897531/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT02897531/ICF_001.pdf